CLINICAL TRIAL: NCT02171351
Title: Effect of Neuromuscular Electrostimulation on Sympathetic Nerve Activity in Patients With Type 2 Diabetes (ELECTROSYMP2)
Acronym: ELECTROSYMP2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issue
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-A00559-38
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2020-08

CONDITIONS: Type 2 Diabetes; Insulin Resistance
Keywords: sympathetic nerve reactivity; neuromuscular electrostimulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- effect of neuromuscular electrostimulation (NMES) (Experimental)
  Interventions: Device: effect of neuromuscular electrostimulation (NMES)
- effect of neuro electrostimulation (NES) (Experimental)
  Interventions: Device: effect of neuro electrostimulation (NES)
- effect of voluntary contractions (VC) (Experimental)
  Interventions: Other: effect of voluntary contractions (VC)

INTERVENTIONS:
Device: effect of neuromuscular electrostimulation (NMES) — Each subject (type 2 diabetes and control) will be assessed with plethysmography during a single session of neuromuscular electrostimulation (NMES).
  Arms: effect of neuromuscular electrostimulation (NMES)
Device: effect of neuro electrostimulation (NES) — Each subject (type 2 diabetes and control) will be assessed with plethysmography during a single session of neuro electrostimulation (NES)
  Arms: effect of neuro electrostimulation (NES)
Other: effect of voluntary contractions (VC) — Each subject (type 2 diabetes and control) will be assessed with plethysmography during a single session of voluntary contractions (VC)
  Arms: effect of voluntary contractions (VC)

SUMMARY:
Physical activity (PA) is recommended for the treatment of subjects with type 2 diabetes to increase insulin sensitivity and improve metabolic control. However, adherence to PA is often poor, due to a lack of motivation or due to disabling complications or comorbidities. Neuromuscular electrostimulation (NMES) is a physical treatment commonly used to improve muscle strength and volume in several situations: after stroke, after limb trauma or during chest rehabilitation in deconditioned patients. The investigators have already shown in a first pilot study (manuscript in preparation) that NMES improves insulin sensitivity : in the study ELECTRODIAB (No. ID-RCB: 2011-A00930-41), the investigators showed a 25% insulin sensitivity improvement after a week of daily 25-min bi-quadricipital NMES session, in a population of patients with orally-treated type 2 diabetes. Insulin sensitivity increased up to 50% in the most deconditioned subjects. Discrepancy between this result and the very low energy expenditure measured during sessions suggests that the metabolic effect was not solely mediated by muscle contractions. The investigators hypothesize the involvement of neurological pathways. Indeed, it is demonstrated that the autonomic nervous system is an important regulator of glucose metabolism with pancreatic action, a key role in energy metabolism and a complex relationship with insulin resistance. Muscle activity, whether static (isometric) or dynamic causes changes in sympathetic nerve activity in healthy subjects but its effect in type 2 diabetic subjects is not known. The investigators hypothesize that, in type 2 diabetic subjects, the modulation of sympathetic nerve activity by NMES could be involved in the improvement of insulin sensitivity. To address this question, the investigators propose to assess sympathetic nerve activity with the gold standard method of microneurography before and after a single bi-quadricipital NMES session. The impact of neuro-electro-stimulation (NES) (a sensitive stimulation under muscular threshold) and the impact of voluntary isometric muscle contractions (VC) will also be evaluated. These procedures will also be applied in healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes for at least 12 month
* treatment by oral hypoglycemic agents and/or GLP1 agonists
* HbA1c : 6-10%
* suspected insulin-resistance (at least one criteria below) :
* waist circumference > 80cm (female); > 94cm (male)
* triglycerides > 150 mg/dl
* HDL-cholesterol < 50 mg/dl (female); < 40 mg/dl (male)
* low background physical activity (Ricci-Gagnon score < 27)

Exclusion Criteria:

* type 1 diabetes
* treatment with insulin
* seizure
* pace maker

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Sympathetic nerve reactivity in response to a single session of neuromuscular electrostimulation | at 0, 5, 10, 15, 20 min of the NMES session
  Sympathetic nerve reactivity will be assessed by plethysmography, with a Valsalva procedure, at baseline and every 5 minutes during a 20-min session of biquadricipital neuromuscular electrostimulation

SECONDARY OUTCOMES:
sympathetic nerve reactivity in response to a single session of neuro electrostimulation | at 0, 5, 10, 15, 20 min of the NES session
  Sympathetic nerve reactivity will be assessed by plethysmography, with a Valsalva procedure, at baseline and every 5 minutes during a 20-min session of biquadricipital neuro electrostimulation
sympathetic nerve reactivity in response to a single session of voluntary muscular contractions | at 0, 5, 10, 15, 20 min of the VC session
  Sympathetic nerve reactivity will be assessed by plethysmography, with a Valsalva procedure, at baseline and every 5 minutes during a 20-min session of biquadricipital voluntary contractions

OTHER OUTCOMES:
comparison of sympathetic nerve reactivity between the different groups and procedures | at 0, 5, 10, 15, 20 min of each session
  sympathetic nerve reactivity will be compared between type 2 diabetic and healthy subjects and between neuromuscular electrostimulation, neuro electrostimulation and voluntary contractions

CONTACTS AND LOCATIONS:
Overall Officials: Michael Joubert, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Clinical Research Center Caen University Hospital, Caen, France